CLINICAL TRIAL: NCT04145245
Title: A Randomized Controlled Trial to Assess the Effect of L-carnitine in Patients With Diabetic Peripheral Neuropathy to Relief Pain and Symptom Improvement
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Farhana Haque, Farhana Haque, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BSMMU/2019/3936
Record Dates: First submitted 2019-10-29; First posted 2019-10-30 (Actual); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Patient Compliance
Keywords: DPN, Levocarnitine
MeSH Terms: conditions — Patient Compliance | interventions — Carnitine

STUDY DESIGN:
Intervention Model Description: Interventional Group- Patients with carnitine in addition to antidiabetic therapy Control Group- Patients with placebo and antidiabetic therapy
Who Masked: Participant, Investigator
Masking Description: placebo controlled, double bind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention or group a (Experimental): Diabetic neuropathy patients with antidiabetic therapy in addition with l-carnitine supplementation
  Interventions: Drug: Levocarnitine
- Placebo or group b (Placebo Comparator): Diabetic neuropathy patients with antidiabetic treatment in addition with placebo
  Interventions: Drug: Levocarnitine

INTERVENTIONS:
Drug: Levocarnitine — Levocarnitine syrup- oral supplementation about 1500 mg/day for 10 weeks
  Other Names: Placebo

SUMMARY:
Diabetic Peripheral Neuropathy (DPN) is a common complication of diabetes mellitus. The prevalence rate is approaching towards a peak throughout the world including Bangladesh. The current intervention used in peripheral neuropathy does not bring satisfactory result. Recent trial shows that L-carnitine is effective and safe in DPN. So it is expected that L-carnitine may produce better effect in compared to other medicine used previously for alleviation of DPN.

DETAILED DESCRIPTION:
: Diabetic peripheral neuropathy is one of the common complication of chronic diabetes mellitus, with a 30-50 % prevalence. Progressive development of pain, numbness in toes or feet and sensory motor disorders affects the patient's quality of life. The epidemic spread of the disease has raised concern among physicians and researchers. A variety of agents or medicines with potential effect have been studied to control development of peripheral neuropathy. The existing management are yet unsatisfactory. Recent studies have suggested that L-carnitine is potential to alleviate symptoms in patents with diabetic neuropathy. Previous trial also indicated the efficacy and safety of L-carnitine on diabetic neuropathy. This limitations have led to search for an effective and tolerable option by placebo controlled trial.The present study is an attempt to investigate the effects of carnitine on pain and symptom improvement of diabetic peripheral neuropathy.

ELIGIBILITY:
Inclusion Criteria:

i. Clinically diagnosed diabetic patients who had been on stable antidiabetic therapy for 1 year ii.Age: 18 years to 70 years iii. Patients HbA1c level <10

Exclusion Criteria:

i. Patient who are suffering from other causes of peripheral neuropathy for example chemotherapy and HIV patient, rheumatoid arthritis, SLE, alcololism, vitamin B12 deficiency etc ii. Lactating and pregnant women iii. Patients taking anticonvulsants, antidepressants, opoioids and other neuropathic pain medication agents

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2018-04-17 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2020-02-28 (Estimated)

PRIMARY OUTCOMES:
VAS score | 10 weeks
  Alleviation of VAS Score of pain

SECONDARY OUTCOMES:
Improvement of neuropathic symptom | 10 weeks
  Alleviation of NSS and NDS of diabetic neuropathy

CONTACTS AND LOCATIONS:
Overall Officials: Farhana Haque, MBBS, Principal Investigator — Resident, phase-B
Locations (1):
- Pharmacology department,BSMMU., Dhaka, Dhaka,Sahbagh, Bangladesh

IPD SHARING:
Plan to Share IPD: No